CLINICAL TRIAL: NCT06195098
Title: A Multidisciplinary and Sustainable Intervention Study Aimed at Rural Area of Madagascar: the Tany Vao Project.
Brief Title: The Tany Vao Project.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: Help for optimism NGO (Unknown); Kukula ONLUS (Unknown); Elpis Nave Ospedale ONLUS (Unknown)
Responsible Party: Principal Investigator, Hellas Cena, University of Pavia, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 04122023
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Malnutrition
Keywords: Malnutrition; Double burden of malnutrition; Sub Saharan Africa; Madagascar; Eating habits; Nutritional knowledge; Nutritional status; Rural areas
MeSH Terms: conditions — Malnutrition; Feeding Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nosy Mitsio Population (Other): Women of childbearing age from 14 to 49 years, pregnant or not and lactating or not, and their children and adolescent form 2 to 18 years old.
  Interventions: Other: Nutritional educational intervention

INTERVENTIONS:
Other: Nutritional educational intervention — The interventional activities were targeted to the local population, according to their educational level and culture and it was composed by a theoretical part and a more practical part. The objective was to improve nutritional knowledge and their awareness about the role of food in connection to the human health. According to the theoretical part: to make the activities more appealing, three informative graphic posters were drafted. According to the practical part: a cooking class activities were conducted, involving women of the Ampanithosa and Bevoko villages. The researchers teaching them how to use a bamboo steamer and how to process vegetables, grew up in the organic gardens built by the Kukula team. The activities were carried out in each village thanks to a local enumerators involvement.

SUMMARY:
The TANY VAO project pilot study aimed to create a circular and sustainable model with a multidimensional and multidisciplinary approach to improve the health conditions of Madagascar's population living in rural areas. This is through an integrated approach in the areas of "wash and sanitation," agriculture, nutrition and "clean cooking." This project consisted of two phases: first an observational phase (Work Package 1, WP1) and secondarily an interventional phase (Work Package 2, WP2). Here is described the nutritional protocol as part of the multidisciplinary study. The nutritional activities were conducted by the Laboratory of Dietetics and Clinical Nutrition (LDNC) of the University of Pavia.

DETAILED DESCRIPTION:
The TANY VAO project pilot study aims to create a circular and sustainable model with a multidimensional and multidisciplinary approach to improve the health conditions of Madagascar's population living in rural areas. This is through an integrated approach in the areas of "wash and sanitation," agriculture, nutrition and "clean cooking."

Here is described the nutritional protocol as part of the multidisciplinary study.

The TANY VAO project was conducted on the island of Nosy Mitsio, 20 miles west of Madagascar, in the villages of Ampanitosoha and Bevoko (western part of the island) on a group of women of childbearing age and their children.

Participants of this study were women of childbearing age (14-49 years old), pregnant or not, and their male or female children/adolescents (2-18 years old) living in the Ampanitosoha and in the Bevoko villages.

Focusing on the nutritional activities the main outcome was to improve food knowledge, eating habits and dietary diversity of the population enrolled in the study.

The project was composed by two different work packages (WP).

WP1: observational phase During this phase researcher were able to catch a picture of the current situation in this specific rural area of Madagascar from a nutritional assessment point of view. Sociodemographic information (religion, civil status, age, educational level) was collected and nutritional knowledge (9-items questionnaire), eating habits (24 hour recall and food frequency), and dietary diversity (minimum dietary diversity index for women) were assessed for women exclusively. A nutritional assessment was conducted for both women and children/adolescents (women: weight, height, abdominal and waist circumference, mid-upper arm circumference, skin fold; children: weight, height, mid-upper arm circumference).

WP2: interventional phase Based on the results of WP1, the interventional activities were defined. The interventional activities were targeted to the local population, according to their educational level and culture and it was composed by a theoretical part and a more practical part. The objective was to improve nutritional knowledge and their awareness about the role of food in connection to the human health. According to the theoretical part: to make the activities more appealing, three informative graphic posters were drafted. The posters provided guidance 1) on food safety and hygiene, 2) on making a complete meal from local foods and practical nutritional advices, and 3) specific indications for the pregnancy and lactation period.

According to the practical part: a cooking class activities were conducted, involving women of the Ampanithosa and Bevoko villages. The researchers taught them how to use a bamboo steamer and how to process vegetables, grew up in the organic gardens built by the Kukula team.

The activities were carried out in each village thanks to a local enumerators involvement.

ELIGIBILITY:
Inclusion Criteria:

* For women: be female, aged between 14 and 49 years and living in the villages of Ampanitosoha and Bevoko (Nosy Mitsio, Madagascar);
* For children/adolescents: male and female subjects, aged between 2 and 18 years; living in the villages of Ampanitosoha and Bevoko (Nosy Mitsio, Madagascar).

Exclusion Criteria:

* Any person who does not fall under the inclusion criteria

Ages: 2 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Improvement of health condition of the study population | 6 months (WP1), 18 months (WP2)
  Nutritional assessment, nutrition knowledge and food intake evaluation, and implementation of nutritional intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, MD, Principal Investigator — University of Pavia
Locations (1):
- University of Pavia, Pavia, Italy

REFERENCES:
- See also: Help for Optimism project description — https://helpforoptimism.org/projects/nutrition-programme/
- See also: Kukula project description — https://kukula.it/tany-vao/